CLINICAL TRIAL: NCT05953922
Title: Effect of Core Stability Exercises on Pain and Quality of Life in Non Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wafaa Ahmed Salama Ashour, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: non specific low back pain
Record Dates: First submitted 2023-05-07; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Non Specific Low Back Pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: intervention study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): The treatment group will engage in transcutaneous electrical stimulation (TENS) and core stability exercises for three sessions each week for four weeks.
  Interventions: Other: core stability exersises
- control group (No Intervention): The transcutaneous electrical stimulation nerve stimulation will be administered to the control group just for three sessions each week for four weeks.

INTERVENTIONS:
Other: core stability exersises — core stability exercises and transcutaneous electrical nerve stimulation for four week three session per week
  Other Names: transcutaneous electrical nerve stimulation
  Arms: treatment group

SUMMARY:
Most publications state that core stability exercises (transverse abdominis and multifidus training) can relieve chronic low back pain with or without radiculopathy and improve function, although only temporarily, and may have the same impact as active general exercise so The goal of this study is to detect the effect of retraining the deep core muscles, on pain, disability, and quality of life in patients with chronic Non specific low back pain.

DETAILED DESCRIPTION:
The goal of this study is to detect the effect of retraining the deep core muscles, on pain, disability, and quality of life in patients with chronic Non specific low back pain

This study is delimited to the following aspects:

1. Fifty, patients of only females with chronic non specific low back pain more than 3 months.
2. The age will range from 22 to 45 years.
3. The treatment will conduct to three session per week for four weeks .
4. The selected patients will assigned randomly to two equal groups:

1- Group1 (intervention), will do the selected treatment that include electrical stimulation in addition to Core stability exercises program. 2- Group2(control), will do the conventional treatment only.

ELIGIBILITY:
Inclusion Criteria:

* gender is women
* age ranges from 22 to45 years old
* chronic non specific low back pain for at least 3 month
* pain score will between 3 to 6 on visual analogue scale

Exclusion Criteria:

* Any deformity of the spine
* Red flags including serious pathology
* Systemic or inflammatory disease
* sever osteoporosis
* history of tumor or cancer
* spine infection
* history of spine or pelvis surgery or fracture
* cauda equina syndrome
* progressive neurological deficit
* severe instability
* sever cardio vascular or metabolic disease
* history of psychological disease
* anatomical and congenital disturbance
* continuous pain more than 8 on (visual analogue scale)

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
quality of life for each participants | baseline
  We will use the Arabic version of world health organization's quality of life (Arabic_WHOQOL-BREF) questionnaire and higher score means better outcome
pain levels for each participants | baseline
  visual analogue scale will be used to assess the level of pain and higher score means worse outcome
pressure lumber biofeedback for each participants | baseline
  pressure lumber biofeedback for asses transverse abdominis contraction

CONTACTS AND LOCATIONS:
Overall Officials: EMAN M. FAYEZ, Professor, Study Chair — Physical Therapy for Neuromuscular Disorder and Its Surgery; Hossam M. Alsaid, Lecturer, Study Chair — Physical Therapy for Neuromuscular Disorder and Its Surgery; MARIHAN Z. Aziz, Lecturer, Study Chair — Physical Therapy for Musculoskeletal Disorders and its Surgery
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Egypt